CLINICAL TRIAL: NCT01921452
Title: A Single-center Interventional Study to Verify Clinical Utility of the Quantitative and the Qualitative POC TSH Test Kits Compared With the Third Generation TSH Test Kit
Brief Title: Study to Verify Clinical Utility of Point-of-Care (POC) Thyroid Stimulating Hormone (TSH) Test Kits as Compared to Third Generation TSH Test Kit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EMR 200125_507
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism; Third generation TSH kit; Quantitative POC TSH kit; Qualitative POC TSH kit
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- POC TSH Kits + Third Generation TSH Kit (Experimental)
  Interventions: Device: Quantitative POC TSH Kit; Device: Qualitative POC TSH Kit; Device: Third generation TSH Kit

INTERVENTIONS:
Device: Quantitative POC TSH Kit — A drop (approximately 30 microliter [mcL]) of blood will be taken from subject's fingertip to test TSH quantitatively by using the quantitative POC TSH test kit according to the product specification on Day 1 to Day 5.
Device: Qualitative POC TSH Kit — A drop (approximately 30 mcL) of blood will be taken from subject's fingertip to test TSH qualitatively by using the qualitative POC TSH test kit according to the product specification on Day 1 to Day 5.
Device: Third generation TSH Kit — One milliliter (mL) of subject's venous blood will be taken to test both qualitative and quantitative TSH levels, by using the third generation TSH test kit on Day 1 to Day 5.

SUMMARY:
This is a Phase 4, single-center, open-label, interventional study, wherein all enrolled subjects will be tested for Thyroid Stimulating Hormone (TSH) by using the quantitative and the qualitative Point-of-Care (POC) TSH test kits and the third generation TSH test kit at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Suspected hypothyroidism subject
* Willing to comply with the trial protocol
* Signed informed consent document

Exclusion Criteria:

* Menstrual period, bleeding hemorrhoids, hematuria
* Drinking or taking aspirin within 48 hours
* Subjects with partially or completely restricted consciousness and behavioral ability, who do not have independent decision-making ability.
* Subjects who are unwilling or unable to complete the trial
* Subjects who do not sign informed consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Limited, UK
Locations (1):
- Research site, Shanghai, China

REFERENCES:
- [Derived] Wang T, Sheng S, Ruan M, Yan J, Gu J, Jiang Y, Gao Y, Lu H. Clinical Evaluation of the Immune Colloidal Gold Method for Rapid Qualitative and Quantitative Measurement of Thyroid-Stimulating Hormone as an Assay for Hypothyroidism. Adv Ther. 2016 Nov;33(11):2001-2011. doi: 10.1007/s12325-016-0401-y. Epub 2016 Sep 7. PMID 27605368

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 283 enrolled participants were analyzed using both point-of-care (POC) thyroid stimulating hormone (TSH) kits and third generation TSH kit.
Groups:
- POC TSH Kits + Third Generation Kit: Participants were analyzed using the following methods on Day 1 to Day 5: (1) POC TSH kits: A drop (approximately 30 microliter [mcL]) of blood was taken from participant's fingertip to test TSH quantitatively and qualitatively by using the quantitative POC TSH test kit and qualitative POC TSH test kit, respectively according to the respective product specifications. (2) Third generation TSH kit: 1 milliliter (mL) of participant's venous blood was taken to test both qualitative and quantitative TSH levels, by using the third generation TSH test kit.
Period: Overall Study
Arm/Group | POC TSH Kits + Third Generation Kit
Started | 283
Completed | 283
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all enrolled participants.
Groups:
- POC TSH Kits + Third Generation TSH Kit: Participants were analyzed using the following methods on Day 1 to Day 5: (1) POC TSH kits: A drop (approximately 30 microliter [mcL]) of blood was taken from participant's fingertip to test TSH quantitatively and qualitatively by using the quantitative POC TSH test kit and qualitative POC TSH test kit, respectively according to the respective product specifications. (2) Third generation TSH kit: 1 milliliter (mL) of participant's venous blood was taken to test both qualitative and quantitative TSH levels, by using the third generation TSH test kit.
Arm/Group | POC TSH Kits + Third Generation TSH Kit
Number analyzed (Participants) | 283
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.99 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181
  Male | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive and Negative TSH Test Result
Time Frame: Day 1 up to Day 5
Population: The FAS included all enrolled participants. 'n' signifies number of participants who were evaluable for this measure for the specified category.
Measure: Number; unit: Participants
Arm/Group | POC TSH Kits + Third Generation TSH Kit
Number analyzed (Participants) | 283
Participants
  POC TSH kits (Positive) (n=282) | 103
  POC TSH kits (Negative) (n=282) | 179
  Third generation kit (Positive) (n=283) | 121
  Third generation kit (Negative) (n=283) | 162

2. Primary Outcome: Concentration of TSH in Whole Blood
Time Frame: Day 1 up to Day 5
Population: The FAS included all enrolled participants.
Measure: Mean (Standard Deviation); unit: Milli international units per liter
Arm/Group | POC TSH Kits + Third Generation Kit
Number analyzed (Participants) | 283
Milli international units per liter
  POC TSH kits | 7.38 (8.49)
  Third generation kit | 30.18 (41.94)

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 5
Description: Safety analysis set included all participants whose blood was collected.
Groups:
- POC TSH Kit + Third Generation TSH Kit: Participants were analyzed using the following methods on Day 1 to Day 5: (1) POC TSH kits: A drop (approximately 30 microliter [mcL]) of blood was taken from participant's fingertip to test TSH quantitatively and qualitatively by using the quantitative POC TSH test kit and qualitative POC TSH test kit, respectively according to the respective product specifications. (2) Third generation TSH kit: 1 milliliter (mL) of participant's venous blood was taken to test both qualitative and quantitative TSH levels, by using the third generation TSH test kit.
Arm/Group | POC TSH Kit + Third Generation TSH Kit
Serious Adverse Events (participants affected / at risk) | 0/283
Other Adverse Events (participants affected / at risk) | 0/283

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review the results communications prior to public release, and the sponsor can embargo communications regarding trial results if the PI does not get approval from the sponsor.